CLINICAL TRIAL: NCT04797325
Title: Open Label Randomized Controlled Clinical Trial of Vedolizumab Versus Conventional Treatment for Checkpoint Inhibitor Induced Colitis
Brief Title: Vedolizumab for Immune Mediated Colitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Emilie Kristine Dahl, Medical Doctor, phd student, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01012121; 2020-005793-10 (EudraCT Number)
Record Dates: First submitted 2021-02-02; First posted 2021-03-15 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Immune-Mediated Colitis
MeSH Terms: interventions — vedolizumab; Prednisolone; Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- vedolizumab (Active Comparator)
  Interventions: Drug: Vedolizumab
- Standard treatment (Active Comparator)
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Vedolizumab — Repeatedly vedolizumab infusion at week 0, 2, 6, 14, 22
  Arms: vedolizumab
Drug: Prednisolone — tablet prednisolone plus infliximab in severe cases.
  Other Names: Infliximab
  Arms: Standard treatment

SUMMARY:
This is an open label randomized trial to evaluate the efficacy and treatment duration with vedolizumab to patients with immune mediated colitis. The trial will include 82 patients randomized into two arms, either standard treatment with prednisolone (plus infliximab in severe cases) or vedolizumab treatment up front.

DETAILED DESCRIPTION:
Background information Immune check point inhibitors (ICPI) have revolutionized the treatment of a growing number of cancer forms resulting in a rapidly increasing number of patients treated with these drugs within the very recent years. The aim is to allow and boost an immune response towards the neoantigens of neoplastic cells, but the blockage of inhibitory signals might also interfere with normal barriers against the development of autoimmunity or autoimmune-like reactions and thus lead to a number of immune-related adverse events (IrAEs). Gastrointestinal inflammation - typically colitis - is the most common IrAE among ICPI treated patients. Vedolizumab, a integrin antibody, has been shown to be highly effective in treating ICPI induced colitis with remission rates of 85%. Vedolizumab has a better safety profile than anti-tumor necrosis factor antibodies, including infliximab, with lower risk of infections and tumor development in inflammatory bowel disease patients. Moreover, vedolizumab does not seem to inhibit tumor specific T cell responses in vitro, suggesting that this treatment is also beneficial with regards to tumor response.

The hypothesis

Vedolizumab induction and maintenance treatment of patients with ICPI related intestinal symptoms and evidence of colitis:

1. Is effective in inducing remission of the colitis
2. Reduces the risk of progression from grade 2 to grade 3 or 4 colitis
3. Reduces the need of systemic corticosteroid
4. Is not associated with increased risk of tumor progression or other serious adverse events including serious infections
5. Allows reintroduction/continuation of ICPI treatment.

Further it is hypothesized that ICPI induced colitis can be diagnosed and monitored by intestinal bowel ultrasound and treatment response is associated with multi-omics changes in intestinal tissue, tumor tissue, feces, blood, and urine, e.g. peripheral blood mononuclear cells (PBMCs) RNAseq profiles, profiles of single cell RNAseq from isolated immune cells from standard pinch biopsies from the inflamed colon and composition of the microbiota. Lastly, it is hypothesized, that anti-tumor T-cell function is affected in vivo by the medication used to treat ICPI induced colitis, and that this can be assessed by changes in single cell RNAseq profiles of tumor resident T-cells (isolated from tumor biopsies).

ELIGIBILITY:
Inclusion Criteria:

* Patients with solid tumors treated with PD-1, PD-L1 and /or CTLA-4 inhibitors and where IrAE colitis is preventing further treatment with check point inhibitors
* IrAE colitis where the oncologist suggests treatment with tablet or IV corticosteroids (prednisolone or equivalent)
* Negative pregnancy test in fertile women
* Age ≥ 18.

Exclusion Criteria:

* Any ongoing infectious disease, including GI infections
* Neutropenia within the last month
* Known allergy towards vedolizumab or Infliximab
* Severe heart failure, NYHA grade 3-4
* Colorectal cancer
* Other IrAEs requiring systemic treatment with either prednisolone (> 10 mg daily or equivalents) or other immunosuppressive medications within 14 days before study drug administration
* Females of childbearing potential or males of reproductive potential who are not willing to use an effective method of contraception, such as oral, injected, or implanted hormonal methods of contraception, intrauterine device or intrauterine system, condom in combination with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam, gel, film, creamer suppository, male sterilization, or true abstinence throughout study and for a minimum of 3 months after study drug therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2021-08-30 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
dose of prednisolone | Week 30
  The cumulative dose of corticosteroids (tablets and IV) due to IrAE colitis at week 30

SECONDARY OUTCOMES:
clinical remission | week 2
  Clinical remission at week 2, 10 and 30*, defined as a partial Mayo score ≤ 2.
clinical remission | week 10
  Clinical remission at week 2, 10 and 30*, defined as a partial Mayo score ≤ 2.
clinical remission | week 30
  Clinical remission at week 2, 10 and 30*, defined as a partial Mayo score ≤ 2.
time to response | 30 days
  Time to clinical remission and eventual relapse of GI symptoms (measured by patient reported stool chart registered the first 30 days).
partial Mayo score | week 2
  Response defined as decrease in partial Mayo score ≥ 30 % at week 2, 10 and 30
partial Mayo score | week 10
  Response defined as decrease in partial Mayo score ≥ 30 % at week 2, 10 and 30
partial Mayo score | week 30
  Response defined as decrease in partial Mayo score ≥ 30 % at week 2, 10 and 30
change in scores | change from week 0 and 10 and 30
  change between clinical scores
fecal calprotectin | change from week 0 and 10 and 30
  change between fecal-calprotectin
IUS | change from week 0 and 10 and 30
  Intestinal ultrasound
endoscopy | change from week 0 and 30
  endoscopy
change in scores | change from week 0 and 10 and 30
  biochemistry
Life qualtity | change from week 0 and 10 and 30
  Changes in quality of life
steroid use for other reasons | During the 30 weeks period
  Corticosteroid use for non-intestinal indications.
ICPI treatment | Week 30
  The proportion of patients able to continue ICPI treatment at any time after inclusion and until week 30*.
steroid free remission | week 10
  Proportion of patients in corticosteroid (tablets or IV) free remission at week 10 and 30* and the cumulative dose corticosteroid at week 10
steroid free remission | week 30
  Proportion of patients in corticosteroid (tablets or IV) free remission at week 10 and 30*
ICPI treatment | week 30
  Proportion of patients able to continue ICPI treatment at any time after inclusion and until week 30

OTHER OUTCOMES:
T-cell response | Change from week 0 to week 15.
  Tumor-specific T cell responses in patients under systemic prednisolone treatment or treatment with infliximab or vedolizumab.
pharmacogenomic | week 0 to week 30
  Pharmacogenomic profiling of genes correlated to ICPI colitis treatment outcome
Omics | week 0 to week 30.
  Omics profiles from blood (buffy coat RNA sequencing transcriptome), urine (metabonome), feces (microbiota, metabonome), and colonic biopsies (RNA sequencing transcriptome)
Single cells | week 0 to week 30
  Single cell RNAseq profiles of PMBCs and single cell RNAseq profiles of immune cells isolated from the mucosal area
Subgroup analysis | week 30
  all outcomes in the subgroup of patients with verified colitis defined as f-calprotectin >200 or endoscopic mayoscore > 0 or intestinal biopsies with evidence of enterocolitis
subgroup analysis | week 30
  all outcomes mentined above in patients without the need of prednisolone during screening

CONTACTS AND LOCATIONS:
Overall Officials: Jakob B Seidelin, professor, Study Director — University of Copenhagen
Locations (1):
- Herlev University Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No